CLINICAL TRIAL: NCT02514642
Title: Safety and Efficacy of Low-dose Ticagrelor in Chinese Patients With Stable Coronary Artery Disease: a Randomized, Single-blind, Crossover Clinical Trial
Brief Title: Safety and Efficacy of Low-dose Ticagrelor in Chinese Patients With Stable Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SCAD-201523
Record Dates: First submitted 2015-07-21; First posted 2015-08-04 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-dose ticagrelor (Experimental): To observe the safety and efficacy of low-dose ticagrelor in Chinese patients withStable Coronary Artery Disease
  Interventions: Drug: low-dose ticagrelor; Drug: Clopidogrel
- clopidogrel (Active Comparator): To observe the different safety and efficacy between low-dose ticagrelor and conventional-dose clopidogrel.
  Interventions: Drug: low-dose ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: low-dose ticagrelor — low-dose ticagrelor (22.5 mg twice daily) for 7 days,followed by a 2-week washout period then a 7days crossover phase of clopidogrel (75mg once daily)
  Other Names: low-dose ticagrelor(22.5 mg twice daily)
Drug: Clopidogrel — clopidogrel (75mg once daily) for 7 days,followed by a 2-week washout period then a 7days crossover phase of low-dose ticagrelor (22.5 mg twice daily)
  Other Names: clopidogrel (75mg once daily)

SUMMARY:
Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy (DAPT) have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for patients who have an ACS with or without ST-segment elevation. However, few East Asian patients (or those of East Asian descent) have been included in these trials to assess the use of these drugs. In Korea and Japan, it has been reported that low doses of ticagrelor might have a more potent inhibition of platelet aggregation (IPA) than clopidogrel (75 mg once daily) in healthy subjects and patients with stable coronary artery disease, respectively. But it is still not clear whether a low dose of ticagrelor is superior to clopidogrel in a large population of Chinese ACS patients. A recent study on pharmacokinetics and tolerability of ticagrelor has found that maximum plasma concentration and area under the plasma concentration-time curve of ticagrelor (90 mg twice daily) and its active metabolite (AR-C124910XX) tended to be approximately 40% higher in healthy Chinese volunteers compared with Caucasian subjects. This data also suggested that a low dose of ticagrelor might be more appropriate for Chinese ACS patients. In view of a large diurnal variation with a single daily dose, a lower dose twice daily may be a better choice for Chinese patients. Therefore, the investigators performed this randomized, single-blind, crossover clinical trial to observe the efficacy and safety of low-dose ticagrelor (22.5 mg twice daily) in comparison to clopidogrel (75mg once daily) in Chinese patients with stable coronary artery disease.

DETAILED DESCRIPTION:
Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy (DAPT) have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for patients who have an ACS with or without ST-segment elevation. However, few East Asian patients (or those of East Asian descent) have been included in these trials to assess the use of these drugs. In addition, a growing body of data supported that East Asian might have different adverse event profiles (thrombophilia and bleeding) and "therapeutic window" compared with white subjects. Furthermore, "East Asian paradox" phenomenon has been also described that East Asian patients have a higher prevalence of platelet reactivity during DAPT, but an ischaemic event rate following percutaneous coronary intervention (PCI) or ACS is similar or even lower than white patients. In Korea and Japan, it has been reported that low doses of ticagrelor might have a more potent inhibition of platelet aggregation (IPA) than clopidogrel (75 mg once daily) in healthy subjects and patients with stable coronary artery disease, respectively. But it is still not clear whether a low dose of ticagrelor is superior to clopidogrel in a large population of Chinese ACS patients. A recent study on pharmacokinetics and tolerability of ticagrelor has found that maximum plasma concentration and area under the plasma concentration-time curve of ticagrelor (90 mg twice daily) and its active metabolite (AR-C124910XX) tended to be approximately 40% higher in healthy Chinese volunteers compared with Caucasian subjects. This data also suggested that a low dose of ticagrelor might be more appropriate for Chinese ACS patients. In view of a large diurnal variation with a single daily dose, a lower dose twice daily may be a better choice for Chinese patients. Therefore, the investigators performed this randomized, single-blind, crossover clinical trial to observe the efficacy and safety of low-dose ticagrelor (22.5 mg twice daily) in comparison to clopidogrel (75mg once daily) in Chinese patients with stable coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Stable Coronary Artery Disease

  1. stable angina
  2. low-risk unstable angina
  3. variant angina
  4. patients with asymptomatic with appropriate therapy（including percutaneous coronary intervention）.

Exclusion Criteria:

1. ACS
2. planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists, or anticoagulant therapy during the study period
3. platelet count <100g/L
4. creatinine clearance rate < 30ml/min
5. diagnosed as respiratory or circulatory instability (cardiac shock, severe congestive heart failure NYHA II-IV or left ventricular ejection fraction < 40%)
6. a history of bleeding tendency
7. aspirin, ticagrelor or clopidogrel allergies
8. diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
P2Y12 reaction units (PRU) | up to 5 months

SECONDARY OUTCOMES:
inhibition of platelet aggregation (IPA) | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, MD, Principal Investigator — Cardiovascular Department, the First Affiliated Hospital of Harbin Medical University
Locations (1):
- VerifyNow, San Diego, California, United States